CLINICAL TRIAL: NCT03173547
Title: A Randomized, Double-blind, Vehicle-controlled Study to Evaluate the Safety and Efficacy of 146-9251 Cream Applied Twice-daily for Six Weeks in Subjects With Ichthyosis Vulgaris
Brief Title: A Six Week Topical Cream Study for Subjects With Ichthyosis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crown Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 146-9251-201
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Ichthyosis Vulgaris
MeSH Terms: conditions — Ichthyosis Vulgaris

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 146-9251 cream (Active Comparator): Topical cream to be applied two times daily to specified treatment areas for 6 weeks.
  Interventions: Drug: 146-9251 cream
- Vehicle cream (Placebo Comparator): Topical cream to be applied two times daily to specified treatment areas for 6 weeks.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: 146-9251 cream — 146-9251 cream contains an active drug and is applied topically.
  Arms: 146-9251 cream
Drug: Vehicle cream — Vehicle cream does not contain an active drug and is applied topically.
  Arms: Vehicle cream

SUMMARY:
The objective of this study is to determine and compare the safety and efficacy of topical 146-9251 cream and vehicle cream applied twice daily for 6 weeks in subjects with moderate to severe ichthyosis vulgaris (IV).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female and is at least 12 years old at the time of enrollment.
2. Subject has provided written informed consent/assent. A subject under 18 years of age must provide written informed assent and be accompanied by the parent or legal guardian at the time of assent/consent signing. The parent or legal guardian must provide informed consent for the subject. If a subject becomes 18 years of age during the study, the subject must provide written informed consent at that time to continue study participation.
3. Subject and parent/guardian (if applicable) are willing and able to apply the test article(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
4. Subject has a clinical diagnosis of ichthyosis vulgaris involving a minimum of 5% body surface area (BSA). If the subject has IV involving over 40% BSA, the investigator must be able to identify a Treatment Area comprising distinct anatomic units that contains about 40% (excluding the scalp and mucosal areas) as detailed in Section 6.2.
5. Subject has an Investigator's Global Assessment (IGA) score of at least three (3 = moderate) at the Baseline Visit.
6. Subject is in good general health and free of any disease state or physical condition that might impair evaluation of IV or which, in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.
7. Females must be post-menopausal, surgically sterile, or use an effective method of birth control. , Women of childbearing potential (WOCBP) must have with a negative urine pregnancy test (UPT) at the Baseline Visit.

Exclusion Criteria:

* 1. Subject is pregnant, lactating, or is planning to become pregnant during the study.

  2. Subject is currently enrolled in an investigational drug or device study. 3. Subject has used an investigational drug or investigational device treatment within 30 days prior to first application of the test article.

  4. Subject has used any topical therapy, including topical corticosteroids or retinoids, in the Treatment Area within 2 weeks prior to the initiation of treatment. Note: a bland emollient may be used in the Treatment Area up to 3 days prior to the initiation of treatment.

  5. Subject has used systemic corticosteroids within 4 weeks or retinoids within 24 weeks prior to the initiation of treatment.

  6. Subject has stable use of vitamin or herbal supplements for less than 2 weeks prior to the initiation of treatment.

  7. Subject has a history of sensitivity to any of the ingredients in the test articles.

  8. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

  9. Subject has a physical condition or other dermatologic disorders (e.g., atopic, seborrheic or contact dermatitis, psoriasis, tinea infections, etc.) which, in the investigator's opinion, might impair evaluation of IV, or which exposes the subject to unacceptable risk by study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Crown investigative site 01, San Diego, California
  - Crown Investigative site 07, Plainfield, Indiana
  - Crown Investigative site 08, Metairie, Louisiana
  - Crown Investigative site 02, Fridley, Minnesota
  - Crown Investigative site 04, Columbia, Missouri
  - Crown Investigative Site 05, Albuquerque, New Mexico
  - Crown Investigative site 06, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 146-9251 Cream | Vehicle Cream
Started | 40 | 40
Completed | 36 | 38
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population defined as subjects who applied at least one dose of the assigned test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | 146-9251 Cream | Vehicle Cream | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (19.41) | 51.4 (17.42) | 53.1 (18.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 21 | 28 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 37 | 37 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 33 | 30 | 63
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Investigator's Global Assessment (IGA) Score [Count of Participants; unit: Participants] — To be eligible for the study, subject must have IGA score of at least three (3=moderate) at their baseline visit.
  Participants
    3-Moderate | 30 | 31 | 61
    4-Severe | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success
Description: Number of participants that show at least a 2 level improvement of overall severity of disease (as measured by IGA score) at 6 weeks. The IGA score is a static evaluation of the overall or "average" degree of severity of a participant's disease, taking into account all of the participant's scaling, erythema, and fissuring in the Treatment Area. IGA was assessed using the following 5-point scale: clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Time Frame: Day 43 (6 weeks)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | 146-9251 Cream | Vehicle Cream
Number analyzed (Participants) | 39 | 39
Participants | 21 | 28

2. Other Pre Specified Outcome: Adverse Events (AEs)
Description: AEs will be assessed by the investigator and the number of participants with any local and systemic AEs will be reported.
Time Frame: Day 0 through study completion, average 6 weeks, Day 43.
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | 146-9251 Cream | Vehicle Cream
Number analyzed (Participants) | 40 | 40
Participants
  Number of Subjects with any AE | 9 | 14
  Number of Subjects without an AE | 31 | 26

ADVERSE EVENTS:
Time Frame: AEs were collected from study day 1 to end of study (week 6).
Arm/Group | 146-9251 Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 5/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 146-9251 Cream (N=40) | Vehicle Cream (N=40)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03173547/Prot_SAP_000.pdf